CLINICAL TRIAL: NCT04906824
Title: Post-Market Registry in Europe and US for the Use of VascuCelTM
Acronym: VascuCel
Status: Active, not recruiting | Type: Observational
Sponsor: LeMaitre Vascular (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Other Study IDs: GLRA-G011
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Great Vessel Reconstruction; Peripheral Vessel Reconstruction; Suture Line Buttressing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: great vessel reconstruction; peripheral vascular reconstruction; suture line buttressing — VascuCel implantation in order to perform great vessel reconstruction; peripheral vascular reconstruction; suture line buttressing

SUMMARY:
This is a post-market, multi-centre, open-label registry designed to collect prospective safety and performance data on the use of VascuCel in patients who require great vessel reconstruction, peripheral vascular reconstruction or suture line buttressing. This registry will collect safety and performance data up to 2 years following implantation.

DETAILED DESCRIPTION:
Post-market, prospective, multi-centre, open-label, registry designed to collect prospective safety and performance data on the use of VascuCel in patients with vascular disorders and in accordance with local standard of care. The Registry has been designed to collect data up to 2 years following implantation. The VascuCel Registry will collect data on the use of the VascuCel, for the following major indications:

* Great vessel reconstruction
* Peripheral vascular reconstruction

As suture line buttressing is a procedure that does not consistently use tissue, data on this indication will only be included if available. Data will be prospectively collected by the sites on registry-specific electronic case report forms (eCRFs). The primary endpoints will assess device's safety and performance through measures and images obtained via the facility's standard of care at the respective registry site. Additional data will also be collected from the implant procedure to assess user (surgeon) satisfaction with the devices' handling and performance.

ELIGIBILITY:
Inclusion Criteria:

* patient has signed the informed consent
* patient is a candidate for treatment with VascuCel per approved device indications.

Exclusion Criteria:

* no study specific exclusion criteria; patients treated per standard clinical practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: VascuCel is indicated for the repair of vascular defects including great vessel reconstruction, peripheral vascular reconstruction and suture line buttressing.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of graft related reintervention | 30 days post procedure.
  collect data on the number of incidence of graft related reintervention
Incidence of patch related morbidity | 30 days post procedure.
  collect data on patch related morbidity

SECONDARY OUTCOMES:
Incidence of graft related reintervention | at 1 and 2 years post procedure.
  collect data on the number of graft related reintervention
Rates of restenosis | at 30 days and 1 and 2 years follow-up
  collect rate of restenosis
Rates of measurement of the dynamic flow by facility standard of care ≥110-175* cm/sec for peripheral vascular location | at 30 days and 1 and 2 years follow-up
  collect rate of measurement of the dynamic flow
incidence of Patch dehiscence | at 30 days and 1 and 2 years follow-up
  collect rate of patch dehiscence
incidence of Patch calcification | at 30 days and 1 and 2 years follow-up
  collect rate of patch calcification
incidence of Patch retraction | at 30 days and 1 and 2 years follow-up
  collect rate of patch retraction
incidence of unanticipated and rare events | at 30 days and 1 and 2 years follow-up
  collect rate of unanticipated and rare events

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Ghiu, Study Director — Anteris
Locations (5):
- United States (4):
  - Kootenai Health, Coeur d'Alene, Idaho
  - Eddy Luh, Las Vegas, Nevada
  - Westchester Medical Center, Valhalla, New York
  - University North Carolina, Chapel Hill, North Carolina
- ASST Sette Laghi Varese, Varese, Italy